CLINICAL TRIAL: NCT00000110
Title: Influence of Diet and Endurance Running on Intramuscular Lipids Measured at 4.1 TESLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Masking: Single | Purpose: Treatment
Other Study IDs: NCRR-M01RR00032-0855; M01RR000032 (NIH)
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Obesity
Keywords: exercise; exertion; physical fitness; lipids; nutrition
MeSH Terms: conditions — Obesity; Motor Activity | interventions — Magnetic Resonance Spectroscopy; Dietary Fats

INTERVENTIONS:
Procedure: magnetic resonance spectroscopy
Drug: dietary fat

SUMMARY:
The purpose of this pilot investigation is to use 1 H Magnetic Resonance Spectroscopy (MRS) to 1) document the change in intra-muscular lipid stores (IML) before and after a prolonged bout of endurance running and, 2) determine the pattern (time course) of IML replenishment following an extremely low-fat diet (10% of energy from fat) and a moderate-fat diet (35% of energy from fat). Specifically, the study will evaluate the change in IML following a 2-hour training run and the recovery of IML in response to the post-exercise low-fat or moderate-fat diet in 10 endurance trained athletes who will consume both diets in a randomly assigned cross-over fashion. We hypothesize that IML will be depleted with prolonged endurance exercise, and that replenishment of IML will be impaired by an extremely low-fat diet compared to a moderate-fat diet. Results of this pilot study will be used to apply for extramural grant support from NIH or the US Armed Forces to investigate the effect of dietary fat on the health and performance of individuals performing heavy physical training. It is anticipated that this methodology could also be employed in obesity research to delineate, longitudinally, the reported cross-sectional relationships among IML stores, insulin resistance and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (developmental phase)
* Healthy endurance-trained subjects
* Maximum age for males is 39
* Maximum age for females is 49

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Alabama at Birmingham Nutrition Sciences Department, Birmingham, Alabama, United States